CLINICAL TRIAL: NCT03436134
Title: Treatment of Chronic Active Antibody Mediated Rejection After Kidney Transplantation by Double-Filtration PlasmaPheresis (DFPP) or Plasma Exchange (PE).
Brief Title: Treatment of Chronic Active Antibody Mediated Rejection After Kidney Transplantation by Double-Filtration PlasmaPheresis or Plasma Exchange
Acronym: DFPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.246
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Kidney Transplantation; Antibody Mediated Rejection
Keywords: Donor-specific antibodies; Double-Filtration PlasmaPheresis (DFPP); Plasma Exchange (PE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma Exchange Group (Active Comparator): Patients receiving Exchange plasma as a treatment of chronic antibody mediated rejection.
  Interventions: Other: Sessions of conventional apheresis
- Double filtration PlasmaPheresis Group (Experimental): Patients receiving double filtration plasmapheresis as a treatment of chronic antibody mediated rejection.
  Interventions: Other: Sessions of news apheresis with double filtration

INTERVENTIONS:
Other: Sessions of conventional apheresis — Patient receiving sessions of Plasma exchange as treatment of chronic antibody mediated rejection.
  The plasma exchange uses a single filter to remove whole plasma and the volume is replaced with a matched volume of blood products +/- saline.) 8 sessions plasma exchange.Patients will have one session per day, 4 consecutive days and then three days without, then one session per day for 4 consecutive days. That's 11 days of treatment at all. The fourth and eighth sessions will be followed by an infusion of Rituximab 375 mg / m2.
  At the beginning and at the end of each session, the patients will have a blood test to measure the parameters of the routine care and the analyzes, collection of biological samples planned for the study.
  Arms: Plasma Exchange Group
Other: Sessions of news apheresis with double filtration — Patient receiving DFPP as treatment of chronic antibody mediated rejection. 8 sessions
  A Double filtration plasmapheresis (DFPP) is a variation of plasma exchange. The circuit contains two plasma filters : the first is a standard plasma filter and the second is a high molecular weight filter that primarily removes immunoglobulins. The depleted plasma is returned to the blood circuit and then to the patient.
  Arms: Double filtration PlasmaPheresis Group

SUMMARY:
In France around 90,000 cases of end-stage chronic kidney disease patients treated either by dialysis (60%) or renal transplantation (just over 40%).

In terms of patient survival and quality of life and also economic reasons, the goal in France is to increase renal transplantation instead of patients on dialysis.

After renal transplant, two main causes of the graft loss after the first years are death of patient with functioning graft, and chronic AntiBody Mediated Rejection (ABMR).

Double Filtration PlasmaPheresis (DFPP) has never been evaluated for this indication.

DFPP makes it possible to treat larger volumes of plasma than plasma exchange, and essentially eliminates higher molecular weights molecules including immunoglobulins comprising DSA (donor-specific alloantibody) but also the C1q involved in the lesions of(ABMR). It is postulated that it will be more effective in treating ABMR than usual plasma exchanges.

A chronic ABMR is the result of the appearance de novo production of anti-Human Leucocyte Antigen antibodies (HLA) against one or more graft antigens (DSA: donor-specific alloantibody).These DSAs will lead to accelerated arteriosclerosis in the graft vessels, which will result in rapidly progressive renal failure, usually associated with a high rate of proteinuria.

Numerous studies have shown that up to 20% of renal transplant patients develop DSA within 5 years of renal transplantation.

Today, no treatment has been shown to be effective in the case of chronic ABMR: the basis of treatment is the reduction/elimination of DSA ( by apheresis for example) and the prevention of its re-synthesis B lymphocytes/plasma cells of the patient (with rituximab for example).

The investigators of this study propose in the context of the active ABMR demonstrated by renal biopsy to evaluate in combination with rituximab, a new apheresis technique double Plasma filtration (DFPP) instead of plasma Exchange.

DETAILED DESCRIPTION:
Each year in the Renal Nephrology and Transplantation Department of Grenoble Hospital treat about twenty renal transplant patients with chronic active antibody rejection. Some patients are diagnosed at a very advanced stage and will not be treated because the expected benefit is tenuous (exclusion criteria).

For both groups, patients will have one session per day, 4 consecutive days then three days without, then one session per day for 4 consecutive days. That's 11 days of treatment in all. The fourth and eighth sessions will be followed by an infusion of Rituximab 375 mg / m2.

At the beginning and at the end of each session, patients will have a blood test to measure the parameters and collection of study biological samples.

DFPP sessions are performed by double filtration technique. A DFPP session lasts about 2 hours for 3.5 L of processed plasma. During the session it is necessary to compensate for 20 grams of albumin.

The plasmapheresis sessions are performed by centrifugation technique. It takes about 20 minutes to prepare the apheresis monitor and circuit. A plasmapheresis session lasts approximately 1h30 for 3.5 L of plasma exchange (replacement with albumin), 2 h for an exchange where the removed plasma is replaced by fresh frozen plasma.

The blood flow rate for plasmapheresis is 80 ml / min, or 50 ml / min a plasma flow rate.

The study includes five follow-up visits following the treatment sessions. A visit 45 days after the start of apheresis sessions, a visit at 3 months and a visit every 3 months for one year.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled into the study, subjects must meet all of the following inclusion criteria

* Kidney transplantation for more than 6 months
* The presence of one or more DSAs with MFI greater than 1000
* Renal Graft dysfunction with renal biopsy of humoral rejection or chronic active antibody mediated rejection lesions based on the 2017 banff score ( with/without C4d)
* Written informed consent in patients

Exclusion Criteria:

Subjects must not be enrolled into the study if they meet any of the following exclusion criteria:

* Kidney transplant for less than 6 months.
* MFI<1000
* Hemoglobin level<110 g/l
* No vascular access patients
* Pre terminal histological lesions of chronic ABMR
* Subject in exclusion period of another study
* Pregnant women, parturient or breastfeeding
* Subject under administrative or judicial control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
show that renal transplant patients with chronic antibody mediated rejection treated with rituximab and DFPP (instead of plasmapheresis +rituximab) had a greater decrease of DSA at 45 days after the end of treatment. | DSA at the first session of the treatment Day1 - At Day 45 post-treatment.
  Measurement of Delta DSA ( evaluated MFI) between Day 45 post-treatment and D0 treatment for every patient in each group

SECONDARY OUTCOMES:
Evaluate of the coagulation parameters (factors II, V, VII, VIII, IX, X, XI, XII, XIII, Von Willebrand and fibrinogen) before/after each session, for each technique (safety) | At day1,day4, day8, day 11, day 45, month 6, month12
  Measurement before/after ratio of factors II,V,VII,VIII,IX,X,XI,XII,XIII,Von Willebrand and fibrinogen in each session for each technique
Evaluate of the serum albumin before/after in each session for each technique (safety) | At day1,day4, day8, day 11, day 45,month 3, month 6, month 9, month12
  Measurement of before/after serum albumin ratio each session and for each technique
Evaluate the complement components C3,C4,C5,C5-9, mannose- binding lectin (MBL) Ficoline3, Properdin and C1q before and after each session for each technique (efficacy) | At day1,day4, day8, day 11, day 45, month 6, month12
  Measurement of ratio before/after complement components ((C3,C4,C5,C5-9, MBL, Ficoline3, Properdin complement and C1q) each session for each technique
Evaluate the immunoglobulin levels(Immunoglobulin G(IgG) , immunoglobulin A: (IgA), immunoglobulin M(IgM)) before and after each session for each technique | At day1,day4, day8, day 11, day 45, month 6, month12
  Measurement of before/after ratio of serum IgG, IgA, IgM in each session for each technique (efficacy)
Evaluate the DSA before the first and after the last session of apheresis in each technique | At day1,day 11, day 45, month 6, month12
  Measurement DSA before the first session and after the last session of apheresis in each technique
Evaluate the following parameters: creatinin, albumin in urine,DSA, levels of MFI, Tacrolimus level. | at Day 0, at day 45, at month 3, at month 9, at month 12
  Measurement serum creatinin level , albumin in urine, creatinin,serum tacrolimus level, DSA, MFI level.
Evaluate renal histological lesions of the chronic antibody mediated rejection at Day45 post-treatment and at Month12 | Biopsy at day45 post treatment. At month 12 post treatment
  pathological analysis of renal biopsy at Day45 and at month12

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Rostaing, PH.MD, Principal Investigator — Nephrology Dialysis Transplantation/ CHU GRENOBLE
Locations (1):
- Grenoble Alpes University Hospital, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eskandary F, Bond G, Kozakowski N, Regele H, Marinova L, Wahrmann M, Kikic Z, Haslacher H, Rasoul-Rockenschaub S, Kaltenecker CC, Konig F, Hidalgo LG, Oberbauer R, Halloran PF, Bohmig GA. Diagnostic Contribution of Donor-Specific Antibody Characteristics to Uncover Late Silent Antibody-Mediated Rejection-Results of a Cross-Sectional Screening Study. Transplantation. 2017 Mar;101(3):631-641. doi: 10.1097/TP.0000000000001195. PMID 27120452
- [Result] Eskandary F, Wahrmann M, Muhlbacher J, Bohmig GA. Complement inhibition as potential new therapy for antibody-mediated rejection. Transpl Int. 2016 Apr;29(4):392-402. doi: 10.1111/tri.12706. Epub 2015 Nov 10. PMID 26474721
- [Result] Gatault P, Kamar N, Buchler M, Colosio C, Bertrand D, Durrbach A, Albano L, Rivalan J, Le Meur Y, Essig M, Bouvier N, Legendre C, Moulin B, Heng AE, Weestel PF, Sayegh J, Charpentier B, Rostaing L, Thervet E, Lebranchu Y. Reduction of Extended-Release Tacrolimus Dose in Low-Immunological-Risk Kidney Transplant Recipients Increases Risk of Rejection and Appearance of Donor-Specific Antibodies: A Randomized Study. Am J Transplant. 2017 May;17(5):1370-1379. doi: 10.1111/ajt.14109. Epub 2017 Jan 3. PMID 27862923
- [Result] Loupy A, Haas M, Solez K, Racusen L, Glotz D, Seron D, Nankivell BJ, Colvin RB, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell L, Drachenberg C, Dragun D, de Kort H, Gibson IW, Kraus ES, Lefaucheur C, Legendre C, Liapis H, Muthukumar T, Nickeleit V, Orandi B, Park W, Rabant M, Randhawa P, Reed EF, Roufosse C, Seshan SV, Sis B, Singh HK, Schinstock C, Tambur A, Zeevi A, Mengel M. The Banff 2015 Kidney Meeting Report: Current Challenges in Rejection Classification and Prospects for Adopting Molecular Pathology. Am J Transplant. 2017 Jan;17(1):28-41. doi: 10.1111/ajt.14107. PMID 27862883
- [Result] Hanafusa N, Kondo Y, Suzuki M, Nakao A, Noiri E, Fujita T. Double filtration plasmapheresis can decrease factor XIII Activity. Ther Apher Dial. 2007 Jun;11(3):165-70. doi: 10.1111/j.1744-9987.2007.00433.x. PMID 17497996